CLINICAL TRIAL: NCT05374811
Title: The Relationship of Neuropathic Pain With Incontinence, Functional Disability and Quality of Life in Patients With Multiple Sclerosis
Brief Title: The Relationship of Neuropathic Pain With Incontinence, Disability and Life Quality in Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Alper mengi, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 26.04.2022/371780
Record Dates: First submitted 2022-05-09; First posted 2022-05-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Disabilities Multiple; Quality of Life; Incontinence, Urinary; Incontinence Bowel; Neuropathic Pain
MeSH Terms: conditions — Multiple Sclerosis; Urinary Incontinence; Encopresis; Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis.: Those diagnosed with Multiple Sclerosis according to the 2017 Revised McDonald criteria
  Interventions: Other: Neuropathic Pain

INTERVENTIONS:
Other: Neuropathic Pain — Neuropathic pain degrees of the patients will be evaluated with the Douleur Neuropathic-4 (DN4) questionnaire.

SUMMARY:
The aim of this study to evaluate the relationship of neuropathic pain with urinary and bowel incontinence, functional disability and quality of life in patients with multiple sclerosis.

DETAILED DESCRIPTION:
The patient's date of birth, gender, education level, body mass index, occupation, marital status, socioeconomic status, who they live with, the onset of their complaints about the disease, the time of diagnosis of multiple sclerosis (MS), the type of MS, the presence of any pain and the type of pain will be recorded.

Then, while the patients will be evaluated by researcher Dr Alper Mengi in terms of neuropathic pain, incotinance, disability and independence in activities of daily living. The forms to be used in terms of health perceptions and quality of life, anxiety and depression, and sleep quality will be filled by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MS according to the 2017 Revised McDonald criteria
* Being between the ages of 18-65
* Being in remission (no progression in attacks or disability in the last 3 months).

Exclusion Criteria:

* Having another known neurological disease
* Having been diagnosed with a psychiatric disease such as depression, anxiety, bipolar disorder
* Having a history of infectious, chronic inflammatory disease, malignancy
* Having cardiac pathology such as heart failure, coronary artery disease
* Diabetes, chronic kidney failure, chronic liver failure
* Being addicted to alcohol and substance
* Using permanent urinary catheter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will consist of patients who applied to the Istanbul University Cerrahpaşa Neurology Multiple sclerosis outpatient clinic between the dates of the study.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Neuropathic pain assessed by Douleur Neuropathic-4 (DN-4) questionnaire. | 7 days
  The patients will be evaluated for neuropathic pain with the Douleur Neuropathic-4 (DN-4) questionnaire. This questionnaire consists of 10 items grouped into four questions: seven items relating to the pain description and to its associated abnormal sensations, and the other three items relating to a brief bedside examination in the painful area. For scoring, 1 is given to each positive and 0 to each negative item. The cut-off value for diagnosis of neuropathic pain is a total score of 4.
Urinary and bowel incotinance assessed by the Functional Independence Measure. | 7 days
  The patients will be evaluated for urinary and bowel incotinance with the sphincter control item of the Functional Independence Measure. Each of the items is graded on a scale of 1-7 based on level of independence in that item (1 = total assistance required, 7 = complete independence).
Disability in multiple sclerosis assessed by the Kurtzke Expanded Disability Status Scale | 3 months
  The patients will be evaluated for disability in multiple sclerosis with The Kurtzke Expanded Disability Status Scale.This scale provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.
Performance in activities of daily living assessed by the Barthel Index. | 3 months
  The patients will be evaluated for performance in activities of daily living with The Barthel Index. The index consists of 10 items that relate to activities of daily living and is calculated by summing the response value to each of these items. The index provides a total score on a scale that ranges from 0 to 100. The Index yields a total score out of 100 - the higher the score, the greater the degree of functional independence.
Health status assessed by Monitoring My Multiple Sclerosis. | 3 months
  The patients with multiple sclerosis will be evaluated for health status with Monitoring My Multiple Sclerosis. This scale consists of 26 items. Answers are evaluated as 1-4 points. The lowest score that can be obtained from the scale is 26, the highest score is 104, and the highest score indicates the satisfaction of the patients with their condition and functions.
The levels of anxiety and depression assessed by Hospital Anxiety and Depression Scale. | 7 days
  The patients will be evaluated for anxiety and depression with Hospital Anxiety and Depression Scale. The scale is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Sleep quality assessed by Pittsburgh Sleep Quality Index. | 1 month
  The patients will be evaluated for sleep quality with the Pittsburgh Sleep Quality Index. It contains 19 self-reported items and 5 items to be completed by a bed partner or roommate, if possible. Scores range from 0 to 3, and are summed to obtain a global score, which ranges from 0 to 21. Higher scores denote greater sleep disturbance.

SECONDARY OUTCOMES:
Descriptive information | 3 months
  The patient's date of birth, gender, education level, body mass index, occupation, marital status, socioeconomic status, who they live with, the onset of their complaints about the disease, the time of diagnosis of multiple sclerosis (MS), the type of MS, the presence of any pain and the type of pain will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Uygunoğlu, MD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)